CLINICAL TRIAL: NCT02112045
Title: A Study of Granix to Disrupt the Bone Marrow Microenvironment in Patients With Multiple Myeloma Undergoing Autologous Stem Cell Transplantation
Brief Title: A Study of Granix to Disrupt the Bone Marrow Microenvironment in Patients With Multiple Myeloma Undergoing Autologous Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to results of interim analysis
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201405057
Record Dates: First submitted 2014-04-04; First posted 2014-04-11 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Filgrastim; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Granix and high dose melphalan (HDM) (Experimental): Granix on Day -7 through Day -2.
  HDM intravenously (IV) on Day -2.
  Autologous stem cell transplantation on Day 0
  Interventions: Drug: Granix; Drug: High dose melphalan (HDR); Procedure: Autologous Stem Cell Transplant (ASCT)
- Control: High dose melphalan (HDM) (Active Comparator): HDM intravenously (IV) on Day -2.
  Autologous stem cell transplantation on Day 0.
  Interventions: Drug: High dose melphalan (HDR); Procedure: Autologous Stem Cell Transplant (ASCT)

INTERVENTIONS:
Drug: Granix
  Other Names: XM02 filgrastim
  Arms: Experimental: Granix and high dose melphalan (HDM)
Drug: High dose melphalan (HDR)
  Other Names: Alkeran® Tablets; Phenylalanine mustard
Procedure: Autologous Stem Cell Transplant (ASCT)

SUMMARY:
This randomized phase II trial compares how well adding XMO2 Filgrastim (Granix) to melphalan before a stem cell transplant works in treating patients with multiple myeloma. Chemotherapy drugs, such as melphalan, are given to prepare the bone marrow for the stem cell transplant. Giving colony-stimulating factors, such as XMO2 Filgrastim (Granix), may help multiple myeloma cells move from the patient's bone marrow to the blood where they may be more sensitive to treatment with melphalan. It is not yet known whether adding XMO2 Filgrastim (Granix) to melphalan before a stem cell transplant will work better than melphalan alone in treating multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma requiring treatment
* Received at least two cycles of any regimen as initial systemic therapy for multiple myeloma and are within 2-12 months of the first dose of initial therapy
* At least 18 years of age
* Adequate autologous stem cell collection, defined as an unmanipulated, cryopreserved, peripheral blood stem cell collection containing at least 2 × 10^6 CD34+ cells/kg based on patient body weight.
* Adequate organ function as measured by:

  * Cardiac function: Left ventricular ejection fraction at rest ≥40%
  * Hepatic function: Bilirubin ≤2 × ULN and aspartate amino transferase/alanine amino transferase (AST/ALT) ≤3 × ULN
  * Renal function: Creatinine clearance ≥40 mL/minute (measured or calculated/estimated)
  * Pulmonary function: Carbon monoxide diffusing capacity (DLCO; corrected for hemoglobin [Hgb]), forced expiratory volume in 1 second (FEV1), forced expiratory vital capacity (FVC) ≥50% of predicted value
  * Oxygen saturation ≥92% on room air
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion Criteria:

* Evidence of multiple myeloma disease progression (as defined by IMWG) any time prior to ASCT
* Prior stem cell transplant (autologous or allogeneic)
* Smoldering MM not requiring therapy
* Plasma cell leukemia
* Systemic amyloid light chain amyloidosis
* Active bacterial, viral, or fungal infection
* Seropositive for human immunodeficiency virus (HIV)
* Known, active hepatitis A, B, or C Infection
* Pregnant or breastfeeding.
* Receiving other concurrent anticancer therapy (including chemotherapy, radiation, hormonal treatment, or immunotherapy, but excluding corticosteroids) within 7 days prior to the ASCT or planning to receive any of these treatments prior to the last study visit on Day +100.
* Hypersensitive or intolerant to any component of the study drug(s) formulation
* Receiving growth factors (filgrastim, XM02-filgrastim, peg-filgrastim, plerixafor, etc) or undergoing apheresis < 14 days prior to the start of treatment on protocol (Day -7).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Jacoby, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 01/20/2015 and closed to participant enrollment on 07/03/2018.
Groups:
- Control: High Dose Melphalan (HDM): HDM intravenously (IV) on Day -2.
Period: Overall Study
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
Started | 45 | 45
Completed | 44 | 45
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM) | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Full Range); unit: years] | 57 [33 to 77] | 62 [40 to 73] | 59.5 [33 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 25 | 43
  Male | 27 | 20 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 45 | 44 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 41 | 38 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response or Stringent Complete Response
Description: Complete response (CR) requires all of the following:
  * Disappearance of monoclonal protein by both protein electrophoresis and immunofixation studies from the blood and urine
  * <5% plasma cells in the bone marrow
  * Disappearance of soft tissue plasmacytomas
  Stringent complete response (sCR) requires all of the following:
  * CR as defined above
  * Normal free light chain ratio
  * Absence of clonal cells in the bone marrow by immunohistochemistry or immunofluorescence
Time Frame: Day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
Number analyzed (Participants) | 44 | 45
Participants | 17 | 17

2. Secondary Outcome: Number of Participants With Adverse Events
Description: -Assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up through Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
Number analyzed (Participants) | 45 | 45
Participants
  Febrile neutropenia | 30 | 27
  Atrial fibrillation | 3 | 2
  Left ventricular systolic function | 0 | 1
  Sinus tachycardia | 1 | 3
  Excessive cerumen | 0 | 1
  Impacted cerumen | 0 | 1
  Dry eye | 0 | 1
  Abdominal pain | 2 | 2
  Colitis | 0 | 1
  Colonic perforation | 0 | 1
  Constipation | 0 | 1
  Diarrhea | 5 | 11
  Enterocolitis | 0 | 1
  Epigastric pain | 0 | 1
  Esophagitis | 0 | 1
  Hemorrhoids | 0 | 2
  Ileus | 0 | 1
  Mucositis oral | 16 | 14
  Nausea | 3 | 5
  Oral pain | 1 | 1
  Upper gastrointestinal hemorrhage | 0 | 1
  Edema limbs | 0 | 1
  Fever | 5 | 4
  Infusion related reaction | 1 | 1
  Malaise | 0 | 1
  Pain | 0 | 1
  Allergic reaction | 1 | 1
  Bacteremia-Coagulase negative staphyococcus | 2 | 1
  Bacteremia - Enterobacter Clocae | 0 | 1
  Bacteremia - Fusobacterium | 0 | 1
  Bacteremia - MSSA | 0 | 1
  Bacteremia - Pseudomonas Aeruginosa | 3 | 1
  Bacteremia - Streptococcus mitis | 1 | 1
  Candida (groin) | 0 | 1
  Clostridium difficile | 3 | 1
  Lung infection | 3 | 3
  Mucosal infection (oral thrush) | 10 | 11
  Peri-rectal yeast infection | 0 | 1
  Sepsis | 1 | 1
  Skin infection | 3 | 3
  Splenic infection | 0 | 1
  Upper respiratory infection | 2 | 4
  Urinary tract infection | 0 | 4
  Vaginal infection | 1 | 1
  Bleeding from CVC insertion site | 0 | 1
  Fall | 2 | 1
  Activated partial thromboplastin time prolonged | 1 | 1
  Aspartate aminotransferase increased | 1 | 1
  Blood bilirubin increased | 3 | 2
  Creatinine increased | 4 | 3
  Electrocardiogram QT corrected interval prolonged | 0 | 1
  Weight loss | 6 | 1
  Anorexia | 1 | 1
  Dehydration | 6 | 3
  Hypernatremia | 1 | 1
  Hyperuricemia | 2 | 1
  Hypoalbuminemia | 18 | 20
  Hypocalcemia | 25 | 22
  Hypokalemia | 16 | 16
  Hyponatremia | 4 | 1
  Hypophosphatemia | 40 | 35
  Bone pain | 4 | 1
  Muscle cramps-back/legs | 0 | 1
  Right thigh/leg pain | 0 | 1
  Acitinic Keratosis (right shoulder) | 0 | 1
  Headache | 1 | 1
  Reversible posterior leukoencephalopathy syndrome | 0 | 1
  Syncope | 0 | 1
  Tremor | 0 | 1
  Anxiety | 0 | 2
  Delirium | 0 | 1
  Insomnia | 0 | 1
  Hematuria | 0 | 1
  Proteinuria | 0 | 2
  Cough | 0 | 1
  Dyspnea | 0 | 1
  Hypoxia | 8 | 5
  Pleural effusion | 0 | 1
  Pulmonary edema | 1 | 1
  Wheezing | 1 | 1
  Erythematous nodules | 0 | 1
  Pruritus | 0 | 2
  Rash acneiform | 2 | 1
  Rash maculo-papular | 0 | 1
  Skin lesion | 0 | 1
  Flushing | 0 | 1
  Hematoma | 0 | 1
  Hypertension | 1 | 1
  Hypotension | 5 | 12
  Phlebitis | 0 | 1
  Thromboembolic event | 3 | 1
  Atrial flutter | 1 | 0
  Myocardial infarction | 1 | 0
  Palpitations | 1 | 0
  Supraventricular tachycardia | 1 | 0
  Adrenal insufficiency | 1 | 0
  SIADH | 1 | 0
  Dyspepsia | 1 | 0
  Dysphagia | 1 | 0
  Hemorrhoidal hemorrhage | 1 | 0
  Odynophagia | 1 | 0
  Chills | 1 | 0
  Multi-organ failure | 1 | 0
  Non-cardiac chest pain | 2 | 0
  Bacteremia - Gram Positive | 1 | 0
  Bacteremia-Serratia liquefaciens/pantoea species | 1 | 0
  Catheter related infection | 1 | 0
  CMV viremia | 1 | 0
  Esophageal infection | 1 | 0
  Otitis media | 1 | 0
  Rhinitis infective | 1 | 0
  Alanine aminotransferase increased | 1 | 0
  Alkaline phosphatase increased | 1 | 0
  INR increased | 3 | 0
  Hyperglycemia | 3 | 0
  Uncontrolled Diabetes Mellitus | 1 | 0
  Generalized muscle weakness | 1 | 0
  Jaw pain | 1 | 0
  Joint effusion | 1 | 0
  Encephalopathy | 1 | 0
  Peripheral sensory neuropathy | 2 | 0
  Presyncope | 1 | 0
  Acute kidney injury | 2 | 0
  Urinary frequency | 1 | 0
  Urinary retention | 1 | 0
  Urinary tract pain | 1 | 0
  Scrotal pain | 1 | 0
  Atelectasis | 1 | 0
  Epistaxis | 1 | 0
  Hiccups | 2 | 0
  Pneumonitis | 2 | 0
  Productive cough | 1 | 0
  Respiratory failure | 1 | 0
  Sore throat | 1 | 0
  Facial rash/dermatitis | 1 | 0
  Follicular rash-back/posterior neck | 1 | 0
  Rash forehead/back | 1 | 0
  Skin ulceration | 1 | 0

3. Secondary Outcome: Number of Participants With Overall Response
Description: Overall response rate=CR+sCR+VGPR+PR
  Complete response (CR), disappearance of monoclonal protein from the blood & urine and <5% plasma cells in bone marrow &disappearance of soft tissue plasmacytomas
  Stringent complete response (sCR), CR & normal free light chain ratio & absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence
  Very good partial response (VGPR), serum and urine monoclonal protein detectable by immunofixation but not on electrophoresis OR > 90% reduction in serum monoclonal protein with urine monoclonal protein < 100 mg per 24 hours and if present, > 50% reduction in the size of soft tissue plasmacytomas
  Partial response (PR), > 50% reduction in the level of the serum monoclonal protein & reduction in urine monoclonal protein & > 50% reduction in the size of soft tissue plasmacytomas & if serum and urine monoclonal protein are unmeasurable and serum free light chain is unmeasurable, a > 50% reduction in plasma cells is required
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
Number analyzed (Participants) | 44 | 45
Participants | 41 | 42

4. Secondary Outcome: Overall Survival as Measured by Number of Participants Alive at Last Follow-up
Description: OS is defined as the duration from the time of transplant Day 0 to death or last follow-up.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
Number analyzed (Participants) | 44 | 45
Participants | 40 | 43
Statistical Analysis 1: Comparison: Experimental: Granix and High Dose Melphalan (HDM) vs Control: High Dose Melphalan (HDM); Test type: Superiority; p = 0.43, Log Rank

5. Secondary Outcome: Progression-free Survival as Measured by Number of Participants Without Disease Progression at Last Follow-up
Description: PFS is defined as the duration from time of transplant Day 0 to time of first progression/clinical relapse, death, or the date the patient was last known to be in remission
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
Number analyzed (Participants) | 44 | 45
Participants | 37 | 36
Statistical Analysis 1: Comparison: Experimental: Granix and High Dose Melphalan (HDM) vs Control: High Dose Melphalan (HDM); Test type: Superiority; p = 0.60, Log Rank

6. Secondary Outcome: Number of Participants With Neutrophil Engraftment
Description: Neutrophil engraftment is defined as ANC ≥ 0.5 × 10^9/L × 3 consecutive daily assessments. The first of 3 consecutive days for which ANC ≥ 0.5 × 109/L will be recorded as the date of neutrophil engraftment. Time to neutrophil engraftment will be calculated as the time from the date of the ASCT to the date of neutrophil engraftment.
Time Frame: Up to Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
Number analyzed (Participants) | 44 | 45
Participants | 44 | 45

7. Secondary Outcome: Number of Participants With Platelet Engraftment
Description: Platelet engraftment is defined as an untransfused platelet measurement >20,000/mm3 × 3 consecutive daily assessments. The first of 3 consecutive days for which the untransfused platelet measurement is >20,000/mm3 will be recorded as the date of platelet engraftment. Time to platelet engraftment will be calculated as the time from receiving the date of ASCT to the date of platelet engraftment. Untransfused is defined as no transfusions within 7 days.
Time Frame: Up to Day 100
Population: 1 participant in control arm did not have a decrease in platelets and is not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
Number analyzed (Participants) | 44 | 44
Participants | 44 | 44

ADVERSE EVENTS:
Time Frame: Reportable adverse events will be collected from the first dose of study treatment (Day -7) through the Day +30 visit.
Description: Reportable adverse events are grade 2 or greater events. Hematologic toxicities are expected and therefore the following adverse events will not be collected or reported regardless of grade: anemia, white blood cell decreased, neutrophil count decreased, lymphocyte count decreased, and platelet count decreased. In addition, the following grade 2 non-hematologic adverse events are expected and will not be reported as adverse events: nausea, vomiting, diarrhea, fatigue, or alopecia.
Arm/Group | Experimental: Granix and High Dose Melphalan (HDM) | Control: High Dose Melphalan (HDM)
All-Cause Mortality (participants affected / at risk) | 40/45 | 43/45
Serious Adverse Events (participants affected / at risk) | 10/45 | 4/45
Other Adverse Events (participants affected / at risk) | 45/45 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Granix and High Dose Melphalan (HDM) (N=45) | Control: High Dose Melphalan (HDM) (N=45)
Atrial filbrillation (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Dehydration (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 3 | 1
Clostridium difficile (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Rhinitis Infective (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Granix and High Dose Melphalan (HDM) (N=45) | Control: High Dose Melphalan (HDM) (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 30 | 27
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Excessive cerumen (Ear and labyrinth disorders) | 0 | 1
Impacted cerumen (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
SIADH (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 11
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Epigastric pain (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 16 | 14
Nausea (Gastrointestinal disorders) | 3 | 5
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Edema limbs (General disorders) | 0 | 1
Fever (General disorders) | 3 | 3
Infusion related reaction (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 1
Bacteremia-Coagulase negative staphylococcus (Infections and infestations) | 2 | 1
Bacteremia-Enterobacter Clocae (Infections and infestations) | 0 | 1
Bacteremia-Fusobacterium (Infections and infestations) | 0 | 1
Bacteremia-Gram positive (Infections and infestations) | 1 | 0
Bacteremia-MSSA (Infections and infestations) | 0 | 1
Bacteremia-Pseudomonas aeruginosa (Infections and infestations) | 3 | 1
Bacteremia-Serratia liquefaciens/pantoea species (Infections and infestations) | 1 | 0
Bacteremia-Streptococcus mitis (Infections and infestations) | 1 | 1
Bleeding from CVC insertion site (Infections and infestations) | 0 | 1
CMV viremia (Infections and infestations) | 1 | 0
Candida (groan) (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0
Clostridium difficile (Infections and infestations) | 2 | 1
Esophageal infection (Infections and infestations) | 1 | 0
Fall (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 1 | 2
Mucosal infection (oral thrush) (Infections and infestations) | 10 | 11
Peri-rectal yeast infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 3 | 3
Splenic infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 0 | 4
Vaginal infection (Infections and infestations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase incrased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 3 | 2
Creatinine increased (Investigations) | 4 | 3
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Hyperglycemia (Investigations) | 3 | 0
INR increased (Investigations) | 3 | 0
Weight loss (Investigations) | 6 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 | 20
Hypocalcemia (Metabolism and nutrition disorders) | 25 | 22
Hypokalemia (Metabolism and nutrition disorders) | 16 | 16
Hyponatremia (Metabolism and nutrition disorders) | 4 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 40 | 35
Muscle cramps-back/legs (Metabolism and nutrition disorders) | 0 | 1
Uncontrolled diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Right thigh/leg pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Actinic Keratosis (right shoulder) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Erythematous nodules (Skin and subcutaneous tissue disorders) | 0 | 1
Facial rash/dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Follicular rash-back/posterior neck (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Rash forehead/back (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 5 | 12
Phlebitis (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT02112045/Prot_SAP_000.pdf